CLINICAL TRIAL: NCT02860871
Title: Use of Infrared Spectroscopy in Septic Arthritis Diagnosis
Acronym: SynoFAST
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC13_8815
Record Dates: First submitted 2016-07-25; First posted 2016-08-09 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-07

CONDITIONS: Joint Effusion
MeSH Terms: conditions — Hydrarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: infrared spectroscopy

SUMMARY:
The main objective of this study is to assess the ability of Fiber-optic Evanescent Wave Spectroscopy (FEWS) to discriminate synovial fluids samples of septic arthritis patients from other causes of joint effusion by analyzing ex vivo joint fluid samples collected during routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* patients benefiting from joint fluid puncture for diagnostic purposes in the rheumatology hospitals participating in the study
* patients over 18 year old,
* patients who received information about the protocol and have not expressed opposition to participate.

Exclusion Criteria:

* patients opposing the study,
* patients aged below 18 year old
* Protected major (safeguard justice , trusteeship and guardianship) and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients benefiting from joint fluid puncture for diagnostic purposes in the rheumatology hospitals participating in the study
Sampling Method: Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of the cause of joint effusion | through study completion, an average of 6 months
  The final diagnosis of the cause of joint effusion is made by the clinician based on the clinical and laboratory data : septic arthritis or other causes of arthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de RENNES, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albert JD, Le Corvec M, Berthoud O, David C, Guennoc X, Hoppe E, Jousse-Joulin S, Le Goff B, Tariel H, Sire O, Jolivet-Gougeon A, Coiffier G, Loreal O. Ruling out septic arthritis risk in a few minutes using mid-infrared spectroscopy in synovial fluids. Rheumatology (Oxford). 2021 Mar 2;60(3):1158-1165. doi: 10.1093/rheumatology/keaa373. PMID 32885254